CLINICAL TRIAL: NCT03441425
Title: Impact of Unexpected Death in Simulation: Skill Retention, Stress and Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20130171-01H
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Crisis Resource Management (CRM) Skills; Stress; Advanced Cardiovascular Life Support (ACLS) Skills
Keywords: CRM Skills; ACLS; Simulation; Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group participants will complete a cardiac arrest simulation scenario on the first day in which the mannequin returns to spontaneous circulation at the end of the scenario. They will then complete a retention simulation session three months later.
- Unexpected death (Experimental): The experimental group participants will complete a cardiac arrest simulation scenario on the first day in which the mannequin unexpectedly dies at the end of the scenario. They will then complete a retention simulation session three months later.
  Interventions: Other: Unexpected death

INTERVENTIONS:
Other: Unexpected death
  Arms: Unexpected death

SUMMARY:
Some educational researchers deliberately induce stress upon learners to in order to enhance retention; this practice is controversial and its utility must be weighed against the negative emotional effects it may have on participants. In this study we investigate the effect of the unexpected death of a simulation mannequin on the retention of non-technical and technical crisis resource management skills and consider the emotional impact of this acute stressor.

DETAILED DESCRIPTION:
Background High-fidelity simulation is an increasingly used teaching tool that is proven to be effective for learning. According to the literature, by gradually increasing stress and emotions, more effective learning can be achieved. However, allowing the simulated patient to "die", as a deliberate stressor, is controversial. There is no previous research on the educational effect of letting a simulated patient die. We aim to evaluate the effects of simulated unexpected death on skill retention, stress levels, and emotions. We hypothesize that the occurrence of unexpected death will impact skill retention, and will be associated with higher stress levels and stronger emotions.

Methods After Institutional Research Ethics Board approval, 56 residents and fellows of different medical specialties will be randomized to either the intervention (unexpected death) or control (survive) group. Participants from both groups will have to individually manage a simulated cardiac arrest crisis. In the intervention group, the scenario will end by the death of the simulated patient, whilst in the control group the simulated patient will survive. Each participant will be immediately debriefed by a trained instructor. Three months later, skill retention will be assessed in a similar scenario. Crisis management performance of all scenarios will be rated by 2 blinded raters. Biological stress, cognitive appraisal, and emotions will be measured during both scenarios.

Implications The impact of simulated unexpected death on skill retention of residents and fellows will provide instructors with evidence to optimize scenario design and approach the role of stress and emotions in simulation-based education.

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident or a fellow in the department of anesthesiology, critical care, emergency medicine, medicine, obstetrics and gynecology, surgery or family medicine at the University of Ottawa or the University of Toronto
* Participants are requested to refrain from physical strains, smoking, drinking caffeinated or low pH beverages and eating for at least one hour before enrollment
* Participants will be included between 11 AM and 8 PM, when cortisol levels are most stable

Exclusion Criteria:

* Not a resident or fellow in one of the departments indicated above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Non-technical Crisis Resource Management (CRM) skills | 3 months
  Assessed using the Ottawa Global Rating Scale

SECONDARY OUTCOMES:
Technical CRM skills | 3 months
  Assessed using a checklist derived from the American Heart Association's Megacode Checklist
Salivary cortisol | 5 time points during each of the 2 simulation days
  Biomarker of stress
State-trait anxiety inventory | 3 time points during each of the 2 simulation days
  Self-perceived anxiety questionnaire
Cognitive appraisal | 2 time points during each of the 2 simulation days
  Ratio of perceived preparedness versus demands of a task
Positive and Negative Affect Schedule (PANAS) | 1 time point during each of the 2 simulation days
  Classification of emotions experienced

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03441425/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03441425/SAP_001.pdf